CLINICAL TRIAL: NCT06396780
Title: Treatment Adherence And Influencing Factors in Children With Helicobacter Pylori Infection During Eradication Therapy: A Cross Sectional Study
Brief Title: Treatment Adherence And Influencing Factors in Children With Helicobacter Pylori Infection During Eradication Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Association Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 039A01
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Helicobacter Pylori Infection; Children, Only
Keywords: H.pylori infection; Medication Adherence; Medication Beliefs; Medication Knowledge; Medication Support; Helicobacter pylori knowledge
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who meet the inclusion/exclusion criteria will be invited to complete the questionnaire: Children will be invited to complete the Medication Adherence Questionnaire, Medication Literacy Questionnaire, and Medication Beliefs Specific Questionnaire. Caregivers will be invited to complete the Helicobacter pylori Knowledge Questionnaire, Medication Beliefs Specific Questionnaire, and Medication Support Questionnaire.

SUMMARY:
The aim of this study is to describe the current status of treatment adherence in children with Helicobacter pylori infection, understand the medication literacy, medication beliefs of the children, knowledge of H. pylori among caregivers, medication beliefs, medication support, and explore the influencing factors of medication adherence.

DETAILED DESCRIPTION:
Helicobacter pylori infection usually occurs in childhood and persists into adulthood, and is closely related to the occurrence of chronic gastritis, peptic ulcer, and gastric cancer. However, in recent years, the eradication success rate of Helicobacter pylori infection has gradually decreased, while the drug resistance rate has gradually increased, and it is urgent to improve the success rate of first eradication in children. Medication compliance is closely related to drug resistance, so it is necessary to investigate medication compliance and its influencing factors during Helicobacter pylori eradication in children.Children and caregivers who meet the inclusion and exclusion criteria were invited to individually complete questionnaire surveys.

Part One: Children infected with Helicobacter pylori and undergoing treatment were invited to complete the questionnaire surveys independently. The children completed the Medication Literacy Questionnaire, Medication Beliefs Specific Questionnaire, and Medication Adherence Questionnaire.

Part Two: Caregivers of the children completed the survey questionnaires, including a demographic information form, H. pylori knowledge questionnaire, Medication Beliefs Specific Questionnaire, and Medication Support Questionnaire.

ELIGIBILITY:
Children Inclusion Criteria:

* 1.Children aged 8-18 years old
* 2. whose diagnosis meets the diagnostic criteria for Helicobacter pylori infection in the Expert Consensus on Diagnosis and Treatment of Helicobacter Pylori Infection in Chinese Children (2022)
* 3. Children who receive Helicobacter pylori eradication therapy

Children Exclusion Criteria:

* 1.Children are diagnosed with other chronic conditions and take other medications for a long time
* 2.Unable to communicate with readers in Chinese normally

Caregiver Inclusion Criteria:

* 1.Caregivers of children who meet the diagnostic criteria for Helicobacter pylori infection in the Expert Consensus on Diagnosis and Treatment of Helicobacter pylori Infection in Children in China (2022)
* 2.Able to communicate normally

Caregiver Exclusion Criteria:

* 1.Not living with children
* 2.Not familiar with the use of children

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eradication of helicobacter pylori in children
Sampling Method: Non-Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Status of adherence | baseline
  Using the Medication Adherence Questionnaire to assess the level of medication adherence in pediatric patients. The questionnaire primarily includes four aspects: adherence to timing, dosage, frequency, and persistence in taking medication. Each aspect consists of four options: (1) Impossible to do; (2) Occasionally possible to do; (3) Basically possible to do; (4) Completely possible to do. Using a scoring method, each option is assigned a score of 1, 2, 3, or 4, respectively, with a score range of 4 to 16 points. Complete adherence is scored as 16 points, basic adherence as 13 to 15 points, minimal adherence as 5 to 12 points, and difficulty as 4 points.

SECONDARY OUTCOMES:
Medication literacy | Baseline
  Medication literacy questionnaire was used to investigate the drug literacy level of children. The questionnaire consisted of 9 items, covering the drug name, dosage and adverse reactions of discharged patients. The 2-point system was used to score points (1 for correct answers and 0 for wrong answers), and the total score of the items was 9 points. Those who scored 0-2 points were considered to have poor drug literacy level, those who scored 3-5 points were considered to have medium drug literacy level, and those who scored 6-7 points were considered to have excellent drug literacy level.
Beliefs about medicine | Baseline
  The Medication Beliefs Specific Questionnaire is used to assess the medication belief levels of pediatric patients and their caregivers. The questionnaire comprises two dimensions: medication necessity and medication concerns, totaling 10 items. Responses are rated on a 5-point Likert scale. Scores for medication necessity and medication concerns dimensions range from 5 to 25 points. Medication belief is calculated as the difference between scores for medication necessity and medication concerns (-20 to 20). Belief levels are categorized as low if the total score is less than 0, moderate if the total score is 0, and high if the total score is greater than 0.
Medication support | Baseline
  The Medication Support Questionnaire assesses caregiver medication support behaviors. The questionnaire consists of 6 items, with each item offering 4 options: ① Impossible to do; ② Occasionally possible to do; ③ Basically possible to do; ④ Completely possible to do. Using a scoring method, each option is assigned a score of 1 to 4 points sequentially. The score range is from 6 to 24 points, with higher scores indicating better caregiver medication support. A score greater than 21 points indicates good caregiver medication support, while a score of 20 or less indicates poor caregiver medication support.
Helicobacter pylori knowledge | Baseline
  Using the Helicobacter pylori Knowledge Questionnaire to investigate the caregivers' level of knowledge about Helicobacter pylori.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol